CLINICAL TRIAL: NCT06924801
Title: Evaluating the Feasibility, Usability, and Integration of the OptiTrack Motion Capture System in Inpatient Physical Therapy
Brief Title: Integration of Real-Time Motion Tracking and Pediatric Rehabilitation
Acronym: Snipperfinger
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 80334
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rehabilitation
Keywords: motion capture technology; Total translational movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patient (Experimental): Pediatric patient will engage with engagement-focused software platform (Snipperfingers) and movement will be analysed by the real-time motion capture system (the OptiTrack system).
  Interventions: Behavioral: Snipperfingers

INTERVENTIONS:
Behavioral: Snipperfingers — Snipperfinger is a self developed engagement focused software platform designed to encourage participation in pediatric physical therapy.

SUMMARY:
Emerging technologies that utilize motion capture integrated with engaging software offer new methods for increasing engagement and movement in patients admitted to the hospital. Hospitalized patients are often limited to sedentary activities, spending the majority of their time in bed, which can contribute to deconditioning and functional mobility deficits. This study seeks to explore the feasibility of a tool designed to promote movement through engaging gameplay that is acceptable to both clinicians and families.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 6-17 years.
* Receiving physical therapy at Stanford Children's Hospital.
* Medically cleared for standing and upper-body movement.
* Ability to follow simple instructions and engage in standing gameplay

Exclusion Criteria:

* Orthopedic or medical conditions contraindicating physical activity.
* Legal guardian not present to obtain consent
* Child with a significant neurological condition or major developmental disability
* Child with active infection of the face or hand
* A history of severe motion sickness A history of seizures caused by flashing light Major surgery within the last 48 hours

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the ease of use of Optitrack system measured by System Usability Scale (SUS) | Post-simulation (5 minutes)]
  10-item questionnaire with a scale from 1- 5, 1 being strongly disagree to 5 being strongly agree on a five-point Likert scale to measure usability.

SECONDARY OUTCOMES:
Acceptability of Intervention Measure (AIM) survey | immediately after the intervention
  This questionnaire consists of 4 items. Measures are to be graded using a 1-5 scale, from 1=completely disagree, to 5= completely agree
Intervention Appropriateness Measure (IAM) survey | immediately after the intervention
  This questionnaire consists of 4 items. Measures are to be graded using a 1-5 scale, from 1=completely disagree, to 5= completely agree
Feasibility of Intervention Measure (FIM) survey | immediately after the intervention
  This questionnaire consists of 4 items. Measures are to be graded using a 1-5 scale, from 1=completely disagree, to 5= completely agree
ISO 9241-400 | immediately after intervention
  6-item ergonomic questionnaire with a scale from 1- 5, 1 being strongly disagree to 5 being strongly agree on a five-point Likert scale.
Setup time required for system use | Before intervention
  Time required to set up the system, defined as the duration from participant arrival in the gym to the start of the physical activity.
Duration of gameplay-driven physical activity | immediately at the start of intervention, immediately after intervention
  Time from first recorded movement in response to gameplay to last movement as recorded by OptiTrack motion capture or clinician observation
Evaluation parent's perception of patient's engagement. | immediately after intervention
  Parent acceptance of the system will be evaluated by self developed questionnaire. The questionnaire contains 10 items with scale from 1-5, 1 being strongly disagree to 5 being strongly agree on a five-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States